CLINICAL TRIAL: NCT00384995
Title: Phase 4 Study of Bicarbonate Versus Saline Infusion Therapy to Prevent Contrast Induced Nephropathy (CAN-IT PREVENT Protocol)
Brief Title: Bicarbonate v Saline to Prevent Contrast Nephropathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Italian Society of Nephrology (Other)
Collaborators: European Commission (Other); Memorial University of Newfoundland (Other)
Responsible Party: Pietro Ravani, Italian Society of Nephrology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR021676
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Kidney Failure, Acute; Contrast Media
Keywords: Contrast Induced Nephropathy; Chronic Kidney Disease; Acute Renal Failure; End-stage Renal Disease; Cardiovascular diseases; Coronary catheterization; Percutaneous coronary intervention; Intra-arterial angiography; Bicarbonate; Saline
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Sodium Chloride; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bicarbonate (Experimental): Bicarbonate solution infusion
  Interventions: Drug: 1/6 M (166 mEq/L) IV Sodium Bicarbonate
- Saline (Active Comparator): Standard volume expansion
  Interventions: Drug: 0.9% (154 mEq/L) IV Sodium Chloride

INTERVENTIONS:
Drug: 0.9% (154 mEq/L) IV Sodium Chloride — Saline solution
  Other Names: Sodium Chloride
  Arms: Saline
Drug: 1/6 M (166 mEq/L) IV Sodium Bicarbonate — Bicarbonate solution
  Other Names: Sodium Bicarbonate
  Arms: Bicarbonate

SUMMARY:
Slowing of kidney function occurs in a minority of people given dye during angiography. The purpose of this study is to compare two different types of fluid given into a vein to reduce the risk of kidney injury: salt in water or baking soda in water.

DETAILED DESCRIPTION:
A decline in kidney function after contrast is associated with prolonged hospital stay, adverse cardiac events, and higher mortality both in hospital and in the long term. Deliberate administration of fluids is recommended to reduce the risk of contrast nephropathy. However, data to support specific recommendations are lacking and the optimal fluid regimen remains unclear.

It has been hypothesized that alkalinization of tubular fluid might be beneficial by reducing pH dependent free radical levels. A recent trial found a lower frequency of creatinine rise > 25% within two days of contrast with a 7 hour infusion of isotonic sodium bicarbonate than with saline infusion (Merten GJ, JAMA 2004). However, it remains to be proven that bicarbonate is superior as this trial has a number of methodological flaws.

Comparison: IV 1/6 M sodium bicarbonate OR IV 0.9% saline, each isotonic fluid given at the same rate of sodium administration (3.25 ml/Kg over 1 hour pre-contrast, followed by 1.1 ml/Kg/hr for 6 hours for bicarbonate; 3.5 ml/Kg over 1 hour pre-contrast, followed by 1.2 ml/Kg/hr for 6 hours for saline). Total infusion time 7 hours (for both). Maximum rate of fluid permitted is that for a body weight of 110 Kg. Intra-vascular iso- or low-osmolality contrast in the minimal dose needed to complete the required imaging.

ELIGIBILITY:
Inclusion Criteria:

* Booked for cardiac or other non-renal arteriography
* Pre-existing reduced kidney function: Serum Creatinine >= 1.3 & <= 4 mg/dl (female gender) or >= 1.5 & <= 5 mg/dl (male gender)
* Age > 18 years

Exclusion Criteria:

* GFR MDRD estimate < 15 ml/min/m2
* End-stage renal disease already on dialysis
* Known current Acute Kidney Failure with serum creatinine rise of > 0.5 mg/dl within 24 hours
* Pulmonary edema - current or within 48 hours
* Clinically relevant ascites, edema or other fluid overload
* Uncontrolled hypertension (> 165 mmHg systolic, or > 105 mmHg diastolic)
* Hemodynamically unstable patient requiring IV nitroglycerine, or IV fluid or inotropes for blood pressure support
* Emergency (unplanned) angiography
* IV contrast procedure
* Exposure to iodinated radiocontrast within 3 days prior to study
* Prior anaphylactoid reaction to contrast
* Planned administration of N-acetylcysteine
* Planned administration of dopamine, fenoldopam or mannitol
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Development of contrast-induced nephropathy, CIN, defined as an increase in serum creatinine of 25% or more from pre-intervention baseline to within 48-72 hours after administration of the radiographic contrast. | 48-72 hours

SECONDARY OUTCOMES:
Group mean change in serum creatinine | 48-72 hours
Days in hospital within the week post contrast | One week
Requirement for dialysis | Two months
Atheroembolic events | Two months
Major adverse cardiovascular events | Two months
Death | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Ravani, MD, MSc, Principal Investigator — Italian Society of Nephrology; Brendan BJ Barrett, MD, MSc, Study Chair — Memorial University of Newfoundland; Ferruccio Conte, MD, Study Chair — Italian Society of Nephrology
Locations (5):
- Italy (5):
  - Spedali Civili di Brescia, Brescia
  - Ospedale Ferrarotto, Catania
  - P.O. Uboldo, Cernusco sul Naviglio
  - Azienda Istituti Ospitalieri di Cremona, Cremona
  - IRCCS Policlinico San Donato, San Donato

REFERENCES:
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Derived] Ravani P, Tripepi G, Pecchini P, Mallamaci F, Malberti F, Zoccali C. Urotensin II is an inverse predictor of death and fatal cardiovascular events in chronic kidney disease. Kidney Int. 2008 Jan;73(1):95-101. doi: 10.1038/sj.ki.5002565. Epub 2007 Oct 17. PMID 17943084